CLINICAL TRIAL: NCT00615667
Title: Prospective, Multicenter Study of the Efficacy and Tolerance of Tacrolimus on Refractory Nephrotic Syndrome (RNS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGNS-001
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Diseases; Nephrotic Syndrome; Tacrolimus
Keywords: Refractory Nephrotic syndrome; Tacrolimus
MeSH Terms: conditions — Kidney Diseases; Nephrotic Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tacrolimus(fk506) treatment (Experimental): tacrolimus(fk506) treatment
  Interventions: Drug: tacrolimus (FK506)

INTERVENTIONS:
Drug: tacrolimus (FK506) — Started: 0.05-0.1mg/kg/d,divided into two daily dose at 12hr; the blood level:5-10ng/ml in induction phase;and 4-6ng/ml in maintenance phase;

SUMMARY:
Exploring the efficacy and safety of Tacrolimus on refractory nephrotic syndrome ; Acquiring the experience of Tacrolimus on the treatment of refractory nephrotic syndrome in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, 14-65 years of age;
2. Diagnosis of Nephrotic syndrome with hypoalbuminemia (<3.0g/dl) and heavy proteinuria (> 3.5g/24hr);
3. Provision of written informed consent by subject or guardian;
4. Refractory nephrotic syndrome:

Steroid resistant: Persistence of proteinuria despite prednisone therapy 1mg/kg/d for 16 weeks; Steroid dependent: NS recurs when steroid dosage decease.Twice within 6 months, and 3 times within 1 year.

Exclusion Criteria:

1. Inability or unwillingness to provide written informed consent ;
2. Known hypersensitivity or contraindication to tacrolimus, cyclophosphamide, azathioprine, corticosteroids;
3. Usage of immunosuppression therapy (MMF, CTX, CysA, MTX ect) for more than 1 week within 1 month prior to first randomization;
4. Pregnancy, nursing or use of a non-reliable method of contraception;
5. Continuous dialysis starting more than 2 weeks before randomization into the induction phase and/or continuous dialysis with an anticipated duration of more than 8 weeks;
6. Previous kidney transplant or planted transplant;
7. Scr > 4mg/dl (353umol/L);
8. Active hepatitis, with liver dysfunction;
9. Diagnosed DM;
10. Participation in another clinic trial and/or receipt of investigational drugs within 4 weeks prior to screening .

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Remission rate | 2006-2008

SECONDARY OUTCOMES:
Renal function, proteinuria, relapse | 2006-2008

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Ping Fu, MD, Principal Investigator — Department of Nephrology, West China Hospital of Sichuan University; Yunhua Liao, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital of Guangxi Medical University; Jin li Zhang, MD, Principal Investigator — Department of nephrology, People's Hospital of Yunnan Province; Jian Chen, MD, Principal Investigator — Department of Nephrology, Fuzhou Military General Hospital; Tanqi Lou, MD, Principal Investigator — Department of Nephrology, 3rd Affiliated Hospital of Sun Yet-Sen University; Yaozhong Kong, MD, Principal Investigator — Department of Nephrology, 1st People's Hospital of Foshan; Junzhou Fu, MD, Principal Investigator — Department of Nephrology,1st People's Hospital of Guangzhou; Wei Shi, MD, Principal Investigator — Department of Nephrology, People's Hospital Guangdong Provincial; Zhengrong Liu, MD, Principal Investigator — Department of Nephrology, Nanfang Hospital of Southern Medical University